CLINICAL TRIAL: NCT00121979
Title: Randomized, Double-Blind, Placebo-Controlled, Multicenter Study Exploring the Safety, Tolerability, and Antiviral Effect of Substituting 600 mg Racivir for 3TC in HIV-Infected Subjects Who Have the M184V Mutation and Are Currently Failing on a HAART Regimen Containing Lamivudine
Brief Title: Study Comparing Racivir and Lamivudine in Treatment-Experienced HIV Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmasset (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CI-PSI-RCV-04-201
Record Dates: First submitted 2005-07-18; First posted 2005-07-21 (Estimated); Last update posted 2007-07-03 (Estimated); Status verified 2005-07

CONDITIONS: HIV Infections
Keywords: HIV; treatment-experienced; lamivudine; 3TC
MeSH Terms: conditions — HIV Infections | interventions — Racivir

INTERVENTIONS:
Drug: Racivir, a non-nucleoside reverse transcriptase inhibitor

SUMMARY:
Racivir ® (RCV) is an experimental drug which means it is not approved for use by the United States Food and Drug Administration (FDA), but it can be used in research studies like this one. RCV (Racivir®) is part of a class of drugs known as "Nucleoside Reverse Transcriptase Inhibitors" (NRTIs), which are intended to block a further increase in the amount of HIV virus in the body. Laboratory research suggests that RCV (Racivir®) may be effective in patients who have developed resistance to other NRTIs, particularly 3TC (lamivudine, Epivir®). However, a study of RCV (Racivir®) has not been done with patients who have previously been treated with other HAART (Highly Active Antiretroviral Therapy -- taking multiple HIV drugs at once) medications including 3TC (lamivudine, Epivir®).

The purpose of this study is to evaluate the safety and effectiveness of RCV (Racivir®) when used together with other HIV drugs in people who have previously been treated with 3TC (lamivudine, Epivir®) and are failing with their current HAART treatments. This study will include a total of 60 HIV infected, HAART-experienced subjects currently receiving 3TC (lamivudine, Epivir®) as part of their HAART therapy. The study will take place at approximately 11 study sites in the US and Latin America.

DETAILED DESCRIPTION:
The study is divided into four periods: a 'Screening' period which can last up to 30 days in duration, a 'Blinded Treatment' period which can last up to 4 weeks in duration, a 'Follow-up' period which is 28 days in duration, and an 'Open-label Treatment' period that some subjects will be given the option to participate in and which can last up to 20 weeks.

If eligible subjects decide to participate in this research study, they will be randomized, which is like picking chances from a hat, to get RCV (Racivir®) alone, 3TC (lamivudine, Epivir®) alone, or RCV and 3TC (lamivudine, Epivir®) in combination. This is a "double-blind study". This means that neither the subject nor the study doctor and study staff will know if subjects are receiving RCV (Racivir®), 3TC (lamivudine, Epivir®), or RCV (Racivir®) and 3TC (lamivudine, Epivir®). This needs to be done to make sure the researchers obtain the information needed to see if RCV (Racivir®) is safe and as effective as 3TC (lamivudine, Epivir®). In case of an emergency, the study doctor will be able to find out immediately what study drug subjects were receiving. With this exception, by signing the consent form subjects agree that they will not be able to find out what medications they are taking, because this is a "double-blind" study, it is necessary to use placebo tablets. A placebo is a tablet that does not contain any active drug, but is made to look just like the study drug.

Subjects will be given three bottles of study medication. They will be asked to take one tablet from each bottle once a day by mouth, in addition to their current HAART drugs, not including 3TC. The 3TC in their current HAART regimen must be discontinued prior to beginning the study medication. It is important that subjects follow all directions when taking the study drugs.

After completing the first 14 days of the blinded treatment period, subjects will be given the option to continue on their current randomized therapy, including their current study medication, for an additional 1-2 weeks. On Day 15, a blood sample will be collected to determine the amount of HIV virus in the blood. Once the results from that blood sample are available, subjects will be told the amount of how much HIV virus changed in the blood during the first 14 days of treatment. Subjects will also be told if they were receiving RCV (Racivir®) alone, 3TC (lamivudine, Epivir®) alone, or a combination of RCV (Racivir®) and 3TC (lamivudine, Epivir®).

If subjects were receiving RCV (Racivir®), to continue in the open-label treatment period, the amount of virus in the blood must drop by at least 2/3 during the first 14 days of the blinded treatment period. For example, if subjects enter the study with 10,000 copies of the HIV virus per milliliter (ml) of blood, then to continue in the open-label period, the virus level must drop to 3,162 copies or less, per ml of blood. Open-label means that participating subjects and the study doctor or study staff will know what treatment subjects were receiving.

If the virus drops by at least 2/3, subjects will be given the option to enter an open-label treatment period. During the open-label period, subjects will receive 600 mg RCV (Racivir®) once daily along with their regular HAART medications. Before entering the open-label period, the study doctor may decide to change the subject's other ARV medications. Participating subjects will be financially responsible for all medications, other than RCV (Racivir®), that the study doctor may prescribe.

Once treatment is "unblinded", subjects may learn that they were not receiving any RCV (Racivir®) during the blinded treatment period. Subjects may voluntarily decide to add 600 mg RCV (Racivir®) once daily to the other HAART medications. The study doctor may decide to change the subject's HAART medications at this time. After 2 weeks of RCV (Racivir®) based treatment, subjects will be asked to return to the study doctor's office to have blood drawn to determine the amount of HIV virus in the blood. Subjects may continue on RCV (Racivir®) for up to an additional 2 weeks until the results from the blood test are available. If the viral load does not decline by at least 2/3, subjects will be withdrawn from the open-label portion of the study. Subjects will be asked to return to the study doctor's office for a final follow-up visit approximately 28 days after the last dose of RCV (Racivir®).

The open-label treatment period will last no longer than 20 weeks. During this study, subjects can receive up to 24 weeks of RCV (Racivir®) therapy. After subjects receive the last dose of study medication, they will enter the follow-up period for 28 days.

If a participating subject or the study doctor decides to withdraw from the study early, subjects will need to return to the study doctor's office to have a follow-up visit approximately 28 days after the last dose of RCV (Racivir®).

ELIGIBILITY:
Inclusion Criteria:

* Males and females who are between 18 years (or the legal age of consent, whichever is older) and 65 years of age. Females may be enrolled following a negative pregnancy test if:

  a) they are documented to be surgically sterile or post-menopausal [amenorrhea >1 year and FSH >30mU/mL]; --OR-- b) they are using a hormonal birth control method (oral contraceptives, contraceptive implants); --OR-- c) they are using a barrier method of contraception (male or female condoms, diaphragm, cervical cap) with a spermicide.
* Subjects with a positive history of HIV-infection, documented by a licensed HIV antibody ELISA assay and confirmed either by Western blot, positive HIV blood culture, positive HIV serum antigen or plasma viremia.
* Subjects currently on an accepted, stable HAART regimen that includes lamivudine for at least 60 days prior to screening.
* Subjects who, in the opinion of the investigator, are failing their current HAART regimen.
* Subjects who have an HIV-RNA copy number of ≥ 2000 copies/mL as determined by FDA-approved, Roche PCR assay (Amplicor HIV-1 Monitor® Test, v1.5 - Quantitative).
* Subjects who have a CD4-lymphocyte count ≥ 50 cells/mm3.
* Subjects who have the M184V HIV mutation, as determined by the FDA-approved Bayer assay, TRUGENE® HIV-1 Genotyping Kit and the OpenGene® DNA Sequencing System.
* Subjects who are able and willing to provide written, informed consent.
* Subjects who are able and willing to comply with the requirements of this study.

Exclusion Criteria:

* Subjects who have a current or recent (< 30 days) opportunistic infection characteristic of AIDS (Category C according to the CDC Classification System for HIV-1 Infection, 1993 Revised Version).
* Subjects currently on a (-)-FTC regimen.
* Subjects with Q151M mutation.
* Subjects with T69S insertions.
* Female subjects who are pregnant or breastfeeding.
* Subjects enrolled in other investigational drug protocols or subjects who have received other investigational agents within 30 days prior to the first dose of study medication. For investigational drugs with an elimination half-life greater than 15 days, this will be extended to 60 days.
* Subjects with malabsorption syndromes possibly affecting drug absorption (e.g. Crohn's disease, chronic pancreatitis, etc).
* Subjects with acute hepatitis B and/or C, except for subjects who, at the discretion of the investigator, have a chronic, but stable hepatitis infection.
* Subjects with the following laboratory parameters within 30 days prior to the first dose of study medication: *Hemoglobin <10.0 g/dL; *Absolute neutrophil count (ANC) <1000/mm3; *Platelet count <100,000/mm3; *AST or ALT >5 times the upper limit of normal, without the presence of an underlying illness, other than HIV or acute hepatitis, judged by the investigator to likely cause such chronic enzyme abnormalities; *Pancreatic amylase >1.5 times the upper limit of normal.
* Subjects who have received an HIV vaccination within 6 months prior to the first dose of study medication.
* Subjects who have received radiation therapy or cytotoxic chemotherapeutic agents within 30 days prior to the first dose of study medication.
* Subjects who, in the opinion of the investigator, are unable to comply with the dosing schedule and protocol evaluations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-09; Study Completion 2006-03

PRIMARY OUTCOMES:
Change from baseline in virological response of HIV (log10 HIV-RNA levels) at the end of week 2
Change from baseline in CD4+ count at the end of week 2
Adverse events

SECONDARY OUTCOMES:
Proportion of subjects in each treatment arm with viral load reduction ≥ 0.5 log10 from baseline
Proportion of subjects in each treatment arm with viral load below 50 copies/mL

CONTACTS AND LOCATIONS:
Overall Officials: Robert Murphy, MD, Study Director — Northwestern University
Locations (6):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - Jacobi Medical Center, The Bronx, New York
  - Burnside Clinic, Columbia, South Carolina
- Fundacion Huesped Clinical Research, Buenos Aires, Argentina
- Instituto Nacional de Nutricion, Mexico City, Mexico
- Medical Research Center Consultorio Royal Center, Republico de Panama, Panama